CLINICAL TRIAL: NCT06678659
Title: A Phase 1 / 2, Open-Label Study of REC-1245 in Participants With Unresectable, Locally Advanced, or Metastatic Cancer
Brief Title: A Study of REC-1245 in Participants With Unresectable, Locally Advanced, or Metastatic Cancer
Acronym: DAHLIA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Recursion Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: REC-1245-101
Record Dates: First submitted 2024-10-29; First posted 2024-11-07 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Unresectable; Locally Advanced; Metastatic Cancers; Relapsed/Refractory Lymphomas
Keywords: RBM39; Cancer; Refractory Lymphomas; Metastatic Cancers
MeSH Terms: conditions — Neoplasms; Lymphoma

STUDY DESIGN:
Intervention Model Description: "Phase 1a: Dose Escalation Phase 1b: Randomized Phase 2: Non-Randomized"
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1a (Experimental): Dose Escalation
  Interventions: Drug: REC-1245
- Phase 1b Dose #1 (Experimental)
  Interventions: Drug: REC-1245
- Phase 1b Dose #2 (Experimental)
  Interventions: Drug: REC-1245
- Phase 2 (Experimental): At recommended Phase 2 dose (RP2D)
  Interventions: Drug: REC-1245

INTERVENTIONS:
Drug: REC-1245 — Oral

SUMMARY:
This is a multi-center, open-label study to investigate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary activity of REC-1245 administered orally on a once daily (QD) schedule in participants with unresectable, locally advanced, or metastatic solid tumors.

DETAILED DESCRIPTION:
Approximately 85 participants will be enrolled in this open-label Phase 1/2 study, allocated 55 participants in Phase 1 and 10-30 participants in Phase 2. The purpose of this study is to investigate the safety, tolerability and pharmacokinetics of REC-1245 for the treatment of participants with unresectable locally advanced or metastatic solid tumors. Participants will receive treatment with REC-1245 for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Have histologically-confirmed unresectable, locally advanced, or metastatic select solid tumors or select relapsed / refractory lymphoma
* Have experienced progressive disease, relapsed disease, or be intolerant to at least one established standard systemic anti-cancer treatment for a given tumor type, or have been considered ineligible for standard therapy.
* Eastern cooperative oncology group (ECOG) performance status ≤ 1
* Measurable disease at baseline per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 / Lugano criteria and documented by computed tomography (CT) and / or magnetic resonance imaging (MRI)

Exclusion Criteria:

* Received treatment with another RBM39 degrader
* Clinically significant gastrointestinal (GI) or GI malabsorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2028-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1-Part 1A (Dose Finding)- Assessment of Dose Limiting Toxicities (DLTs) | Initiation of study drug through 4 weeks
  To characterize the incidence of DLTs
Phase 1 and 2 -Treatment-emergent Adverse Events | Initiation of study drug through 30 days after the last dose (up to approximately 24 months)
  To characterize the incidence of treatment emergent adverse events
Phase 2- Objective Response Rate (ORR) | Initiation from study drug until disease progression (up to approximately 24 months)
  To assess tumor response

SECONDARY OUTCOMES:
Phase 1- ORR | Initiation from study drug until disease progression (up to approximately 24 months)
  To assess tumor response
Phase 1 and 2- Disease Control Rate (DCR) | Initiation from study drug until disease progression as applicable (up to approximately 24 months)
  To assess the anti-tumor activity
Phase 1 and 2 - Duration of Response (DOR) | Initiation from study drug until disease progression as applicable (up to approximately 24 months)
  To assess the anti-tumor activity
Phase 1 and 2 - Duration of Stable Disease (SD) | Initiation from study drug until disease progression as applicable (up to approximately 24 months)
  To assess the anti-tumor activity
Phase 1 and 2 - Time to Response (TTR) | Initiation from study drug until disease progression as applicable (up to approximately 24 months)
  To assess the anti-tumor activity
Phase 1 and 2 - Progression Free Survival (PFS) | Initiation from study drug until disease progression as applicable (up to approximately 24 months)
  To assess the anti-tumor activity
Phase 1 and 2 - Overall Survival (OS) | Initiation from study drug until disease progression as applicable (up to approximately 24 months)
  To assess the anti-tumor activity
Phase 1 - Maximum Plasma Concentration (Cmax) | Initiation of study drug through Week 9
  To characterize PK of REC-1245
Phase 1 - Time to Reach Maximum Plasma Concentration (Tmax) | Initiation of study drug through Week 9
  To characterize PK of REC-1245
Phase 1 - Plasma Concentration Before the Next Dose (Ctrough) | Initiation of study drug through Week 9
  To characterize PK of REC-1245
Phase 1 - Area Under Plasma Concentration-time Curve (AUC) | Initiation of study drug through Week 9
  To characterize PK of REC-1245

CONTACTS AND LOCATIONS:
Locations (6):
- United States (4):
  - City of Hope, Duarte, California
  - Cleveland Clinic, Cleveland, Ohio
  - SCRI Oncology Partners - PPDS, Nashville, Tennessee
  - START Mountain Region, West Valley City, Utah
- Canada (2):
  - McGill University Health Centre (MUHC) - The Montreal, Québec, Canada
  - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No